CLINICAL TRIAL: NCT05387187
Title: Evaluate the Effect and Safety of Pu Yang Wan Wu Tang and Western Medicine on Chronic Kidney Disease
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Su, Po-Hsuan, Principal Investigator, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N202204011
Record Dates: First submitted 2022-05-11; First posted 2022-05-24 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pu Yang Wan Wu Tang plus Pentoxifylline (Experimental)
  Interventions: Drug: Pu Yang Wan Wu Tang plus Pentoxifylline
- Pentoxifylline (Active Comparator)
  Interventions: Drug: Pentoxifylline

INTERVENTIONS:
Drug: Pu Yang Wan Wu Tang plus Pentoxifylline — Pu Yang Wan Wu Tang 5g TID Pentoxifylline 100mg TID
  Arms: Pu Yang Wan Wu Tang plus Pentoxifylline
Drug: Pentoxifylline — Pentoxifylline 100mg TID
  Arms: Pentoxifylline

SUMMARY:
The indication of Pu Yang Wan Wu Tang is stroke sequelae, such as half body paralysis, aphasia and muscle weakness.

Pu Yang Wan Wu Tang is proved to have the effect of protecting nerve and blood vessel, anti-inflammation, anti-coagulation, dilating peripheral vessel, promot-ing micro circulation, improving hemodynamics, and activating central nerve system. Huangqi could attenuate podocyte injury by regulating the expression and distribu-tion of nephrin and podocin. Huangqi and Danggui are associated with fewer infiltra-tion of macrophages and limitation of renal intrinsic cell activation, which may lead to earlier and persistent reduction of proteinuria.

This research will use the compound Chinese medicine, Pu Yang Wan Wu Tang. Those treatments combined Western medicine to assess the efficacy and drug safety on the CKD cases. Series of blood and urine were collected regularly during study to prove the role of Chinese medicine in the treatment of CKD, and to assess their drug safety.

The final goal of the plan is to establish the new indication of Pu Yang Wan Wu Tang and enhance the interaction and cooperation between Chinese and Western medicine.

ELIGIBILITY:
Inclusion Criteria:

* Participants' age is between 20 to 80 years.
* Participants CKD stage are from 2 to 4(eGFR from 89 to 15)
* Participants under regular western medicine therapy.
* Participants who agree to follow the trial protocol.
* Participants who can complete the study treatment and assessments.

Exclusion Criteria:

* Participants who are already under hemodialysis, Peritoneal Dialysis or kidney transplant.
* Participants who are participating in other clinical trials.
* Participants with hematopoietic system diseases, severe psychiatric or psychological disorder, or cancer.
* Women who are pregnant.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Value of eGFR | At baseline
Value of eGFR | At 4-weeks
Value of eGFR | At 8-weeks
Value of eGFR | At 12-weeks

SECONDARY OUTCOMES:
Value of Creatinine | At baseline
Value of Creatinine | At 4-weeks
Value of Creatinine | At 8-weeks
Value of Creatinine | At 12-weeks
Value of BUN | At baseline
Value of BUN | At 4-weeks
Value of BUN | At 8-weeks
Value of BUN | At 12-weeks
Ratio of Urine Protein/Urine Creatinine | At baseline
Ratio of Urine Protein/Urine Creatinine | At 4-weeks
Ratio of Urine Protein/Urine Creatinine | At 8-weeks
Ratio of Urine Protein/Urine Creatinine | At 12-weeks
Value of GOT | At baseline
Value of GOT | At 4-weeks
Value of GOT | At 8-weeks
Value of GOT | At 12-weeks
Value of GPT | At baseline
Value of GPT | At 4-weeks
Value of GPT | At 8-weeks
Value of GPT | At 12-weeks

CONTACTS AND LOCATIONS:
Overall Officials: PO-HSUAN SU, MD, Principal Investigator — Taipei Medical University Hospital
Locations (1):
- Taipei Medical University, Taipei, Taiwan